CLINICAL TRIAL: NCT06049966
Title: Effectiveness of Atezolizumab in Large Cell Neuroendocrine Carcinoma of the Lung and the Value of miR21 and miR-375 as Biomarkers
Brief Title: Atezolizumab in Large Cell Neuroendocrine Carcinoma
Acronym: LANCE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncology Center of Biochemical Education And Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPI-2023-2304
Record Dates: First submitted 2023-09-10; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Large Cell Neuroendocrine Carcinoma of the Lung
Keywords: Atezolizumab; Immunotherapy; LCNEC; Large Cell Neuroendocrine Carcinoma; Immune Checkpoint Inhibitors; miR375
MeSH Terms: interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Carboplatin 5 AUC D1 plus Etoposide 100mg/m2 D1-D3 plus Atezolizumab 1200 mg, Q21, 4 Cycles and then maintenance Atezolizumab 1200 mg Q21
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Arm B (Active Comparator): Carboplatin 5 AUC D1 plus Etoposide 100mg/m2 D1-D3, 4 Cycles and then observation
  Interventions: Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Atezolizumab — TECENTRIQ C/S.SOL.IN 1200MG/VIAL (20ML) 1 VIAL x 20ML
  Other Names: Tecentriq
  Arms: Arm A
Drug: Carboplatin — SOL.INF 450MG/45ML VIAL ΒΤx1VIALx45ML
  Other Names: CARBOPLATIN/HOSPIRA
Drug: Etoposide — ETOPOSIDE/PHARMACHEMIE SOL.INF 100MG/5ML VIAL BT x 10 VIALS x 5 ML

SUMMARY:
Large Cell Neuroendocrine Carcinoma (LCNEC) is a rare and aggressive form of cancer that presents significant challenges regarding treatment options and prognosis. In this trial, the effectiveness of Atezolizumab in treating metastatic LCNEC was evaluated. Atezolizumab is an anti-PD-L1 antibody that has shown promising results in other types of cancer, such as small-cell lung Cancer and non-small-cell lung cancer. The trial aimed to assess the efficacy and safety of atezolizumab in combination with chemotherapy as a potential treatment option for treatment-naive patients with metastatic LCNEC The trial was conducted as an open-label, non-randomized study, comparing Atezolizumab plus platinum etoposide to platinum etoposide alone in patients with metastatic LCNEC.

DETAILED DESCRIPTION:
This trial is a prospective clinical study to evaluate the effectiveness of a combination treatment regimen for patients with metastatic Large Cell Neuroendocrine Carcinoma (LCNEC) originating from the lung. The trial occurred between March 2018 and August 2022 at the 3rd Department of Medicine, Kapodistrian Medical School of Athens. The institutional review board of Sotiria Chest Diseases Hospital of Athens approved it. The trial adhered to Good Clinical Practice guidelines and the Declaration of Helsinki, and all patients or their legal representatives provided informed consent.

Patients:

The trial enrolled patients with metastatic LCNEC originating from the lung. Eligible patients had not received prior systemic treatment for LCNEC. Patients with brain metastases at diagnosis underwent Whole Brain Radiotherapy (WBRT) before starting systemic treatment.

Study Design:

The experimental group received a combination treatment regimen consisting of four cycles of Carboplatin, Etoposide, and Atezolizumab every 21 days.

Patients who achieved stable disease (SD) or a response (partial or complete) continued maintenance treatment with Atezolizumab until disease progression or discontinuation due to severe adverse events.

The control group received four cycles of Carboplatin and Etoposide. Immune checkpoint inhibitors were not allowed in later lines of treatment for the control group.

Response to therapy was assessed using CT scans and physical evaluations.

Endpoints:

Progression Free Survival (PFS): The time from treatment initiation to disease progression or death.

Overall Survival (OS): The time from treatment initiation to death. Overall Response Rate (ORR): The percentage of patients with a complete or partial response based on RECIST v1.1 criteria.

Duration of Response (DoR): The length of time the disease responded to treatment without progression on imaging studies.

Procedure:

Patients were treated at the 3rd Department of Medicine, Kapodistrian Medical School of Athens.

Approval for immunotherapy was obtained from the National Organisation for the Provision of Health Services (EOPYY) for each patient.

Blood samples for miR-375 and miR-21 analysis were collected at specific time points and processed according to standard procedures.

Analysis of miRNA expression was performed using the miRCURY LNA SYBR Green PCR Kit.

Statistical Analysis:

Rstudio was used for statistical analysis. The trial did not include a power analysis. The intention-to-treat principle was followed. Kaplan-Meier methods and Cox Regression survival analysis were used to estimate PFS and OS.

An analysis of the significance of the difference in characteristics between the experimental and control groups was conducted.

miR-21 and miR-375 Analysis:

Control samples for miR-21 and miR-375 were collected from volunteers without a cancer diagnosis, matching age with LCNEC patients.

Blood samples were collected at specific time points and processed to isolate plasma.

RNA was isolated from plasma samples, followed by cDNA synthesis and miRNA quantification using the miRCURY LNA SYBR Green PCR Kit.

MiR-103a-3p was used as a reference gene. Real-time PCR was performed to quantify miRNAs, and the results were expressed relative to the control group.

ELIGIBILITY:
Cohorts A and B:

Inclusion Criteria:

* Histologically confirmed Stage IV (metastatic) or unresectable locally advanced LCNEC
* No prior treatment
* With or without brain metastasis, if symptomatic patients should be treated with WBRT first
* Performance Status ≤ 2
* Life expectancy > 3 months
* Written informed consent
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

Exclusion Criteria:

* Prior treatment with chemotherapy, immunotherapy, targeted small molecule therapy, or radiation therapy (except WBRT for brain metastasis from LCNEC)
* Active or history of autoimmune disease or immune deficiency
* Treatment with systemic immunosuppressive medications with the following exceptions:

Patients who have received acute, low-dose systemic immunosuppressant medication (≤ 10 mg/day oral prednisone or equivalent) or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained.

* Major surgical procedure other than for diagnosis within 4 weeks before initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Active malignancy or malignancy within 3 years
* Active tuberculosis
* Current severe, uncontrolled systemic disease other than cancer
* Known clinically significant liver disease
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, an average of 3 years
  Progression Free Survival (PFS) was defined as the time from treatment initiation to disease progression οr death. Patients alive without progression at the last follow-up were censored at the date of the deadline for follow-up
Overall survival | Through study completion, an average of 3 years
  Overall survival (OS) was defined as the time from treatment initiation to death, and patients alive during the last follow-up were censored at the date of the deadline for follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N Syrigos, Study Chair — National and Kapodistrian University of Athens; Georgios Evangelou, Principal Investigator — National and Kapodistrian University of Athens; Konstantinos N Syrigos, Study Director — Konstantinos
Locations (2):
- Greece (2):
  - National and Kapodistrian University of Athens, Athens
  - OCEBER, Athens

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF